CLINICAL TRIAL: NCT02926040
Title: Impact of Irreversible Electroporation on Quality of Life for Patients With Locally Advanced Pancreatic Cancer
Brief Title: Quality of Life After in Situ IRE in Locally Advanced Pancreatic Cancer
Acronym: IRE Qol
Status: Terminated | Type: Observational
Why Stopped: PI left hospital
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: St. Claraspital AG (Other); Cantonal Hospital of St. Gallen (Other); Cantonal Hospital of Zug (Unknown)
Responsible Party: Sponsor
Other Study IDs: KEK 2016-01458
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Irreversible electroporation

SUMMARY:
A. Pancreatic cancer background In 2012, 1,172 new pancreatic cancer patients were diagnosed in Switzerland. Only 20% of the patients with newly diagnosed pancreatic cancer are candidates for surgical resection, the only potential treatment for cure. Over 30% of the patients initially present with locally advanced disease. Patients with locally advanced disease have no evidence of metastatic spread to the liver, lung, and peritoneum but present with local involvement of vital structures that prohibits reasonable tumor resection. Currently, those patients are evaluated for palliative chemotherapy +/- radiation therapy. However, even with best conventional medical therapy, median survival of patients with locally advanced disease is mostly below 1 year. Over the last years, loco-regional therapies gained increased attention including radiofrequency-, cryo-, and microwave ablation as well as electrochemotherapy. However, all those entities are criticized by their complication rates leading to morbidity and mortality, limited area of application given the complex anatomical structures around the pancreas, and ill-defined improvements in overall survival.

B. Irreversible electroporation (IRE):

Irreversible electroporation is an emerging ablative modality that gained enormous interest over the last five years. For locally advanced pancreatic cancer, it was introduced in 2009. IRE is mainly non-thermal and primarily works through apoptosis. Its well studied safety profile allows ablation also within the context of locally advanced pancreatic cancer given it mainly spares vessels from destruction.

Increasing evidence shows that IRE for locally advanced, unresectable pancreatic cancer is effective compared to historic controls with a significant prolongation of local progression free survival, distant progression free survival and overall survival. The improvement in overall survival is about double the amount of what is seen with best new chemotherapy and chemoradiation regimens used at the present time. Those results are even more impressive given the discouraging improvements among palliative systemic options.

The NanoKnife IRE device (Angiodynamics, Queensbury, NY) is commonly used to perform IRE procedures in pancreatic cancer patients and is commercially available since 2009 and got Food and Drug Administration (FDA) 510K clearance for soft tissue ablation in October 2011 in the United States.

C. Quality of life and nutritional status/long term outcomes Given the overall poor long-term outcomes of patients with pancreatic cancer, health-related quality of life (HRQoL) measures are of utmost importance when treatment recommendations are discussed with patients. This is especially true for patients with more advanced staged disease where definitive surgical resection with curative intent is not possible. However, HRQoL reports for patients with locally advanced pancreatic cancer undergoing IRE are very limited. To the best of the investigators' knowledge, no other specific investigations exist that assessed HRQoL measures for patients undergoing IRE for locally advanced pancreatic cancer, no specific assessment exists that focuses on nutritional status for this patient group. In addition, impact on local and distant recurrence as well as cancer-specific and overall survival are still ill-defined and further information is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to undergo general anesthesia (ASA ≤3)
* Performance status ECOG <=2 (Eastern Cooperative Oncology Group)
* Locally advanced, unresectable, histology proven pancreatic adenocarcinoma
* Partial response or stable disease after a minimum of 3 months of (radio-) chemotherapy after diagnosis of pancreatic adenocarcinoma without signs of liver or lung metastases
* Last chemo-/radiotherapy procedure >4 weeks ago

Exclusion Criteria:

* Cardiac conduction abnormalities (e.g. AV-conduction abnormalities)
* History of epilepsy
* Recent history of myocardial infarction (2 months)
* Metallic biliary stent that is not removable prior to procedure by endoscopy and within the ablation field
* Evidence of distant metastasis (e.g. liver, lung, peritoneum)
* Informed consent cannot be given by the patient
* Known hypersensitivity to the IRE electrodes (stainless steel 304L)
* Women of childbearing potential who are pregnant, breast feeding, or not taking an adequate method of contraception at the time of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HRQol measured by health questionnaire | day 7
  Quality of life health questionnaire
Change from baseline in HRQol measured by health questionnaire | day 21
  Quality of life health questionnaire
Change from baseline in HRQol measured by health questionnaire | day 42
  Quality of life health questionnaire
Change from baseline in HRQol measured by health questionnaire | day 90
  Quality of life health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Worni, MD, Principal Investigator — Inselspital
Locations (3):
- Switzerland (3):
  - Clarahospital, Basel
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Zug, Zug